CLINICAL TRIAL: NCT01179945
Title: Effects of a Food Preservative on Glucose Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 10-05-0202
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Overweight
Keywords: diabetes; benzoic acid; benzoate; soda; soft drink; preservative; blood sugar
MeSH Terms: conditions — Overweight; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- sodium benzoate containing (Experimental)
  Interventions: Other: benzoate containing test drinks
- non sodium benzoate containing (Active Comparator)
  Interventions: Other: non sodium benzoate containing test drinks

INTERVENTIONS:
Other: benzoate containing test drinks — Subjects will consume 500ml of water with 0.5 grams of sodium benzoate, followed by a solution of 75g sugar in 500ml water with 0.5 grams sodium benzoate 3 hours later.
  Each solution will be consumed over 5 minutes.
  Arms: sodium benzoate containing
Other: non sodium benzoate containing test drinks — Subjects will consume 500ml of water followed by a solution of 75g sugar in 500ml water 3 hours later.
  Each solution will be consumed over 5 minutes.
  Arms: non sodium benzoate containing

SUMMARY:
The investigators propose to examine the effects of the common food preservative sodium benzoate on blood glucose and related hormones and metabolites. If an effect is demonstrated, patients with increased diabetes risk could be counseled to avoid this preservative.

DETAILED DESCRIPTION:
Soft drink consumption has been repeatedly implicated in the development of type 2 diabetes (T2DM). Interestingly, epidemiology studies have yielded inconsistent results. Some studies identify sugar-sweetened beverages as the culprit, whereas others point towards artificially-sweetened beverages. Beyond differences in methodology, these conflicting reports raise the question whether another ingredient common to both sugar and artificially-sweetened soft drinks, such as a preservative, might play a role.

Benzoate salts are widely used preservatives in products such as sodas, canned goods, and pharmaceuticals. Interestingly, there is published evidence that sodium benzoate and its metabolite hippurate can affect pancreatic islet function and impair glucose tolerance. However, the effects of oral sodium benzoate at concentrations typically used in our diet on glucose homeostasis have not been systematically studied. Here, we propose to close this knowledge gap.

We will recruit 15 healthy, overweight volunteers, age 18-35. Each subject will receive 4 interventions: an oral glucose challenge 1) with and 2) without 0.1% benzoic acid, and a drink of water 3) with and 4) without 0.1% benzoic acid. Blood samples will be analyzed for glucose, insulin, glucagon, and a panel of approximately 300 different metabolites at baseline and serially for 2 hours after each intervention. Factorial analysis of variance will be performed to determine the effects of benzoic acid in the presence and absence of glucose, and interactions between glucose and benzoate. The planned sample size of 15 will provide 80% power to detect an effect-size of 0.16 standard-deviations in outcome measures, and an interaction-effect of 0.33 standard-deviations, with a critical value p=0.05.

If we find through this study that sodium benzoate significantly affects glucose tolerance, the public health implications would be great. High level, frequent consumption might cause diseases associated with insulin resistance, chiefly T2DM. Furthermore, its presence in OGTT testing solutions could provide misleading results.

ELIGIBILITY:
Inclusion Criteria:

* Men and women age 18-35
* BMI 25-30

Exclusion Criteria:

* Diabetes Mellitus (fasting Blood Glucose ≥ 126mg/dl)
* Exercise more than 60 minutes more that 4 times a week
* Major medical illness
* Medications or supplements that can influence glucose metabolism
* Large fluctuations in weight (>5% over the past 6 months)
* Currently following a weight loss program
* Consumption of more than 24 ounces of soda per day (defined as sugar- or artificially sweetened beverages, e.g. colas or fruit punches, excluding hot tea and coffee)
* Allergy or intolerance to sodium benzoate
* Nicotine use
* Illicit substance use
* Women with irregular menstrual cycles, or who are pregnant or breastfeeding

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2010-08; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Blood glucose area under the curve (AUC) | 120 minutes post ingestion
  Plasma glucose will be measured at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution, and area under the curve will be calculated.

SECONDARY OUTCOMES:
Insulin AUC | 120 minutes
  Serum Insulin will be measured at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution, and area under the curve will be calculated.
Glucagon AUC | 120 minutes
  Plasma Glucagon will be measured at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution, and area under the curve will be calculated.
Metabolite Profiles | 120 minutes
  Metabolite analysis will be performed on blood samples at baseline, 15, 30, 45, 60, 90, and 120 minutes post ingestion of each test solution, and area under the curve will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: David S Ludwig, MD, PhD, Principal Investigator — Boston Children's Hospital; Vamsi Mootha, MD, Principal Investigator — Massachusetts General Hospital; Belinda S Lennerz, MD, PhD, Study Director — Boston Children's Hospital; Scott Vafai, MD, Study Director — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts